CLINICAL TRIAL: NCT03320811
Title: Interpretation of Serological Tests in the Diagnosis of Celiac Disease: Anti-deamidated Gliadin Peptide Antibodies Revisited
Acronym: DGP-CeliacDis
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2016Ao005
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Celiac Disease
Keywords: Celiac disease; serological tests; anti-deamidated gliadin peptide antibodies
MeSH Terms: conditions — Celiac Disease | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group "celiac disease"
  Interventions: Other: Data record
- group "no celiac disease"
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record

SUMMARY:
Celiac disease is an autoimmune disorder characterized by a chronic inflammation of the small bowel mucosa, triggered by the ingestion of gluten-containing grains.

The diagnosis of celiac disease was initially based on duodenal biopsies obtained from upper endoscopy. Since 1990, the availability of serological tests has contributed to a different perception of the disease. Serological testing is now considered fundamental for celiac disease screening, even if duodenal biopsies remain the gold standard. Celiac markers usually include anti-TG2 antibodies, anti-endomysium antibodies, anti-gliadin antibodies and anti-reticulin antibodies. Recently, several studies showed that deamidated products of gliadin may enhance T-cell stimulatory activity and improve the reactivity of anti-gliadin antibodies. Thus, detection of anti-deamidated gliadin peptide antibodies has been introduced into the wide spectrum of serological tests for celiac disease.

DETAILED DESCRIPTION:
The aim was to assess the clinical relevance of anti-deamidated gliadin peptide antibodies compared with the other common celiac markers.

ELIGIBILITY:
Inclusion Criteria:

- patients attending the Reims University Hospitals, for whom serological tests for celiac disease were prescribed between 1 april 2012 to 31 december 2014

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients attending the Reims University Hospitals, for whom serological tests for celiac disease were prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 2026 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
celiac disease | Day 0
  The celiac disease diagnosis was based on the histological lesions at duodenal biopsies (villous atrophy). Biopsy samples were obtained during upper gastrointestinal tract endoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France